CLINICAL TRIAL: NCT04468789
Title: Evaluation of the National Department of Health's Six-month Antiretroviral Treatment Dispensing Demonstration Pilot in Primary Health Care Clinics in the Context of the COVID-19 Pandemic and Response in South Africa
Brief Title: Evaluation of Six-month HIV Treatment Dispensing in South Africa
Status: Withdrawn | Type: Observational
Why Stopped: The South African government decided not to implement the pilot project for which this protocol was the evaluation. It was not approved by the IRB and never started.
Sponsor: Boston University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Other Study IDs: H-40512; OPP1192640 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2021-05

CONDITIONS: HIV
Keywords: HIV; antiretroviral therapy; multi-month dispensing; South Africa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Comparison group: Patients eligible for six-month dispensing receiving care at comparison sites.
- Intervention group: Patients eligible for six-month dispensing receiving care at intervention sites.
  Interventions: Other: Six-month ARV dispensing

INTERVENTIONS:
Other: Six-month ARV dispensing — Patients in the intervention group who meet eligibility criteria will receive a six-month supply of antiretroviral medications, rather than the standard of care supply which is typically 2-3 months.
  Groups: Intervention group

SUMMARY:
Many countries in sub-Saharan Africa are implementing a policy of six-month dispensing of antiretroviral (ARV) medications for HIV. Under the new guidelines, stable patients can receive a six-month supply of ARV medications at once, reducing the number of clinic visits required for medication refills. South Africa is considering this policy but has not yet adopted it and has requested evidence of its feasibility, effectiveness, and costs to the healthcare system and to patients. The decision on whether to implement a six-month dispensing policy has become urgent due to the SARS-Cov-2 epidemic, as clinic visits to refill prescriptions pose COVID-19 transmission risks to both patients and providers.

To generate the required evidence, South Africa is implementing a pilot program that will allow for a cluster-randomized evaluation of 6-month dispensing. This protocol is for that evaluation. It aims to provide supporting evidence to inform future policy and procurement decisions by the National Department of Health (NDOH). All interventions will be conducted as part of routine care by Department of Health staff.

In the pilot program, the NDOH will randomize 28 clinics in two provinces 1:1 to receive the six month dispensing intervention or continue standard of care, which currently allows for 2-3 month dispensing. The researchers will assess the patient outcomes of six month dispensing, administer a cross-sectional patient questionnaire, conduct semi-structured in-depth interviews with care providers and implementers, and estimate the costs to NDOH and to patients of six month dispensing. A maximum of 150,545 patients will be followed through their medical records and 400 patients and providers will be consented to be interviewed at baseline and after 6 months (total maximum sample size = 150,945).

DETAILED DESCRIPTION:
The overall aims of this study are to assess the uptake and impact of six-month medication dispensing (6MMD) on HIV patients' treatment outcomes at public-sector clinics; estimate the costs of the intervention; and assess patients' and providers' perspectives on 6MMD. All implementation of the interventions and generation of data will be done by the National Department of Health and its support partners; this study will evaluate the outcomes.

The specific objectives of the evaluation are to:

Objective 1: Among HIV infected patients on antiretroviral therapy who are newly eligible for 6MMD, assess the uptake of 6MMD among eligible patients, stratified by repeat prescription refill strategy. Evaluation questions:

* What proportion of patients is eligible for 6MMD?
* What proportion of eligible patients choose to enrol in 6MMD?
* What proportion of enrolled patients receive more than one consecutive 6-month refill?

Objective 2: Is six-month dispensing non-inferior to standard of care (two- or three-month dispensing) in terms of retention in care and viral suppression? Evaluation questions:

* What is the effect of 6MMD on retention compared to standard of care for patients eligible for 6MMD?
* What is the effect of 6MMD on viral suppression within 6 and 12 months of intervention enrollment (intervention patients) or eligibility (comparison patients), compared to standard of care for patients eligible for 6MMD?
* What is the effect of 6MMD on retention and suppression among all ART patients in a clinic, regardless of whether they were eligible for or received 6MMD?

Objective 3: Is 6MMD more or less acceptable to patients and providers than standard of care? Evaluation questions:

* What factors influence patient choice to enrol in 6MMD?
* To what extent does the risk of COVID-19 influence a patient's decision to enrol in 6MMD?
* What are the barriers and facilitators to implementing 6MMD from the perspective of providers?
* How has COVID-19 impacted the implementation of 6MMD?
* Has there been any task shifting as a result of the implementation of 6MMD?
* What was the level of fidelity to the standard operating procedures (SOP) for 6MMD implementation?

Objective 4: What is the cost of 6MMD to providers and patients compared to standard of care. Evaluation questions:

* How often do 6MMD patients return to facilities for HIV or other health care or to collect other chronic medications between scheduled ARV dispensing visits?
* What is the average cost to the provider (DOH) per 6MMD patient and for all ART patients at the study clinics?
* What is the patient cost of ART for those receiving 6MMD compared to standard of care?

ELIGIBILITY:
Inclusion Criteria:

* Objectives 1 and 2: On same ART treatment regimen for at least 6 months; most recent viral load taken in the past 6 months; and last viral load undetectable (<50 copies/ml3)
* Objective 3: Patient at an intervention site who meets the eligibility criteria for 6MMD; or provider at an intervention site

Exclusion Criteria:

* Objectives 1 and 2: Not resident in the facility's catchment area; recorded intention to transfer care to a different facility within 12 months; or pregnant and eligible for PMTCT
* Objective 3: Not resident in the facility's catchment area; recorded intention to transfer care to a different facility within 12 months; pregnant and eligible for PMTCT; unable to communicate in one of the language into which the consent documents and questionnaire have been translated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Objective 1: All adult, HIV-positive patients who have initiated antiretroviral therapy at the study sites Objective 2: All adult, HIV-positive patients who have initiated antiretroviral therapy at the study sites Objective 3: Adult, HIV-positive adults eligible for six-month dispensing at the intervention sites; and providers at the intervention sites
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Uptake of 6MMD | Baseline
  Proportion of patients eligible for 6 multi-month dispensing (6MMD) who enroll in 6MMD at intervention sites
Retention in care | 6 months
  Proportion of patients eligible for 6MMD who are retained in care at 6 months
Viral suppression | 12 months
  Proportion of patients eligible for 6MMD who are virally suppressed at 12 months

SECONDARY OUTCOMES:
Provider acceptability of 6MMD before intervention | Baseline
  Acceptability of 6MMD to healthcare providers, based on interview responses
Provider acceptability of 6MMD after intervention | 6 months
  Acceptability of 6MMD to healthcare providers, based on interview responses
Patient acceptability at baseline | Baseline
  Acceptability of 6MMD to patients, based on survey responses
Patient acceptability at 6 months | 6 months
  Acceptability of 6MMD to patients, based on survey responses
Provider costs | 12-months
  Costs to healthcare provider (study clinics) of 6MMD, compared to standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Rosen, Principal Investigator — Boston University
Locations (1):
- Health Economics and Epidemiology Research Office, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No